CLINICAL TRIAL: NCT01006239
Title: The Biorepository for Scripps Health
Acronym: BIF
Status: Active, not recruiting | Type: Observational
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Principal Investigator, Eric Topol, MD, Director, Scripps Translational Science Institute, Scripps Translational Science Institute
Other Study IDs: IRB 09-5261
Record Dates: First submitted 2009-10-29; First posted 2009-11-02 (Estimated); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Cancer
Keywords: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will be collecting solid tumor and adjacent non-diseased tissue from patients undergoing surgical resection of a solid tumor.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Biorepository: Patients undergoing surgical resection of a solid tumor.
  Interventions: Other: No study intervention

INTERVENTIONS:
Other: No study intervention — The is no study related intervention.

SUMMARY:
The investigators propose to establish a Biorepository of both diseased and normal tissue collected from subjects undergoing surgery for solid tumor resection. In cooperation with the Scripps Cancer registry, the investigators will also establish an anonymized database of corresponding clinical information including response to treatment, disease status, and recurrence.

The Biorepository for Scripps Health will be able to process, preserve, and distribute samples to scientific and medical researchers at Scripps.

DETAILED DESCRIPTION:
Biorepository samples will be utilized in a variety of research studies intended to help in the diagnosis and/or treatment of patients, including the possible identification of therapeutic targets or genetic identifiers of cancers and possibly other diseases. Various technologies including gene expression, genotyping, DNA and RNA sequencing, protein and metabolite analysis may be used in the course of the various studies An exemplary project currently under consideration is one in which Scripps Genomic Medicine is comparing the DNA sequence of both a patient's tumor and their germline DNA to identify genetic differences between the two. These differences could help identify specific pathways that are regulating the tumor and disease thus leading to potentially valuable information in how to treat that individual patient as well as other patients with similar genetic characteristics. In addition, differences between the tumor and germ-line observed in multiple patients could help identify therapeutic targets that are cancer specific. A secondary exemplary project which is currently underway is one in which Scripps Genomic Medicine is undertaking RNA sequencing to identify "fusion genes" which are hybrid genes formed from two previously separate genes and are a type of genetic mutation that has been identified in certain types of cancers including those of the prostate and breast and certain forms of leukemia. Identifying new fusion genes could provide valuable insights into both treatment protocols and new therapeutic targets.

The goal of this project is to expand and improve the bio-repository already established within the Scripps Genomic Medicine (SGM) group. Presently, the collection has been focused on the collection of predominately prostate tumors and blood as the corresponding normal tissue. The current collection is annotated with pathology information and limited medical information collected from the patient during the consenting process; no post surgical information is collected. We believe that collection can be enhanced by (i) modifying the tumor collection process, (ii) simplifying the means of consenting the patients such that it relies upon the general surgical consent and (iii) using de-identified medical data already consolidated in the Cancer registry as a means of annotating the tissue samples.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Undergoing surgical resection of solid tumor
* Completion of general surgical consent (authorizing "pathologist to use his or her discretion in the disposition or use of any tissues removed during surgery or other procedure unless otherwise directed by my physician. I understand that tissues that are removed may be used for teaching purposes as well as research, institutional or commercial".)

Exclusion Criteria:

* Does not meet all of the inclusion criteria above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects over the age of 18 undergoing surgical resection of solid tumor.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2009-11; Primary Completion 2025-12 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Establish a Biorepository of both diseased and normal tissue | six years
  Establish a Biorepository of both diseased and normal tissue

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Topol, MD, Principal Investigator — Scripps Translational Science Institute and Genomic Medicine
Locations (1):
- Scripps Mercy Hospital, San Diego, California, United States